CLINICAL TRIAL: NCT00971958
Title: Infant Male Circumcision in Gaborone, Botswana, and Surrounding Areas: Feasibility, Safety and Acceptability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rebeca Milanesi Plank, MD, Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2007p-002142
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; Circumcision
Keywords: HIV prevention; infant, neonatal, male circumcision
MeSH Terms: conditions — HIV Infections | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mogen Clamp (Active Comparator)
  Interventions: Procedure: Circumcision; Device: Mogen Clamp; Device: Plastibell; Device: AccuCirc
- Plastibell (Active Comparator)
  Interventions: Procedure: Circumcision; Device: Plastibell; Device: AccuCirc
- AccuCirc (Active Comparator): AccuCirc is a device approved by the FDA for circumcision of male infants up to ten days of life.
  Interventions: Device: Plastibell; Device: AccuCirc

INTERVENTIONS:
Procedure: Circumcision — Neonatal circumcision using one of three non-experimental, widely available devices.
  Arms: Mogen Clamp; Plastibell
Device: Mogen Clamp — Mogen clamp is a reusable, one-size stainless steel clamp use for neonatal circumcision.
  Arms: Mogen Clamp
Device: Plastibell — The plastibell is a one-time use device for the circumcision of male neonates, infants and children.
Device: AccuCirc — AccuCirc is a device used for the circumcision of male infants approved for use by the FDA up to 10 days of life.

SUMMARY:
Background: Novel HIV prevention approaches are urgently needed in Botswana and elsewhere in sub-Saharan Africa. Although adult male circumcision (MC) has been shown to reduce the heterosexual acquisition of HIV by men by about 60%, MC in infancy is optimal for its relative ease, lower cost and low rate of complications. We have conducted focus groups and semi-structured interviews that suggest neonatal MC (< 28 days of life) would be an acceptable public HIV prevention strategy in Botswana. The government of Botswana is committed to scaling up MC services in the immediate future and they plan to include neonates. Understanding decision-making around infant MC will be essential to maximize the effectiveness of this HIV prevention strategy.

Specific Aims: The investigators propose to: 1) determine the acceptability and actual uptake of neonatal MC in southeastern Botswana and identify barriers to uptake; 2) ascertain the feasibility and safety of neonatal MC in Botswana; 3) Estimate what, if any, advantages would exist for scale up of Mogen Clamp, Plastibell or AccuCirc with regard to human resources, equipment needs, adverse events and acceptability to health-care providers and families in Botswana.

Study Design and Schema: The investigators will conduct structured interviews with early postpartum mothers and fathers to determine correlates of neonatal MC acceptability and uptake, defined as neonatal MC following informed consent. Male infants will be circumcised by a trained doctor in a hospital / clinic setting by one of three FDA-approved devices that are currently in use in US hospitals: Mogen clamp, Plastibell or AccuCirc. Circumcision with Mogen Clamp or Plastibell will be done before 29 days of life. Circumcision with AccuCirc will be done before 11 days of life (FDA approval limit for device). The investigators will also administer questionnaires to the parents at the regular pediatric follow-up visit(s) to assess impressions of / satisfaction with the infant's procedure outcome over time. Provider impressions of the three methods will also be evaluated. Sample size will be 150 infants per arm for a total of 450 infants males circumcised (and an estimated 800 parental questionnaires).

Public Health Significance: The World Health Organization (WHO) and UNAIDS state that countries with severe, generalized HIV epidemics but low rates of MC should offer this surgery as an important, evidence-based HIV prevention intervention, including among neonates. These two agencies also recommended that additional research on the most feasible, safe, and sustainable ways of scaling up MC intervention should be performed. This study will be in keeping with these recommendations.

Please note the Mogen clamp and Plastibell study arms began as a randomized trial before the initiation of the AccuCirc single-arm portion. Although the settings in which the three devices were studied were similar, the AccuCirc trial enrollment began at two sites (Gaborone and Molepolole) only after completion of the Mogen clamp and Plastibell arms, which was conducted in three sites (Gaborone, Molepolole and Mochudi). Although Lobatse was a site for the first acceptability study with mothers, no procedures were performed there.

Regarding the reported sample size: the total, final sample size includes both parents of newborn boys (because enrolled consenting parents completed questionnaires as part of this study), and boys whose parents consented to circumcision. We anticipated that not all parents who completed the questionnaire would consent to circumcising their baby; therefore, when planning the study it was necessary to estimate the number of parents who would participate in the survey (700), to achieve an enrollment of 300 neonates (therefore the initial estimate of 1000). The original study in fact enrolled 302 infants, 600 mothers and 19 fathers (total study population 921). The addition of the AccuCirc arm led to a revised estimate of total number of neonates and their parents (total=1250). The final enrollment was of 1,235 participants, that includes all the participating neonates and parents.

ELIGIBILITY:
Inclusion Criteria:

* Mothers (and fathers) of liveborn male infants at one of the four study sites who are > 21 years of age (mothers less than 21 years of age, age of majority in Botswana, will provide assent, and will need consent from a guardian to allow participation of mother and infant in this study).
* Fathers of liveborn male infants at one of the four study sites who are > 21 years of age
* Ability to follow up regularly at study clinic until 4 months postpartum
* Provision of written informed consent

Exclusion Criteria:

* Neonatal sepsis or other severe illness requiring infant hospitalization
* Penile abnormality that might require reconstructive surgery in the future (penile torsion / median raphe not midline, hypospadias / blind urethral pit, buried penis, penile-scrotal web, hydrocoele, dorsal hood / ventral foreskin missing, lack of scrotal ruggae suggesting lack of testicles bilaterally as could be karyotypic XX, megameatus or any other abnormality that may require consultation with urologist)
* Family history of bleeding disorder
* Estimated infant gestational age < 37 weeks
* Infant delivery weight < 2,500 grams
* Infant > 4 weeks of age
* Infant receipt of methaemoglobin-inducing agents
* Current involuntary incarceration of mother

Max Age: 28 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1235 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Adverse events that were potentially related to neonatal MC were defined prior to study initiation and categorized as bleeding, infection, structural and other. | Within 6 weeks
  Bleeding requiring only the application of pressure beyond the immediate post-procedure period was defined as a minor adverse event. Intervention other than pressure (e.g. suturing) was defined as a moderate adverse event. A separate clinic visit or hospitalization for bleeding from the circumcision site or need for IV fluids or blood products were categorized as major adverse events. Infection limited to the circumcision site was defined as a minor adverse event. Soft-tissue infection spreading beyond the penis (lower abdominal wall, upper legs) was defined as a moderate adverse event. Systemic infection / sepsis was defined as a major adverse event. Removal of too much or incorrect tissue; removal of too little tissue requiring repeat procedure; or structural injury to glans, urethra or shaft were defined as major adverse events, as were subsequent problems with urination or proximal migration / retention of a Plastibell ring requiring intervention for removal.
Parental Satisfaction | At 6 weeks and 4 months
  As to parental satisfaction, we asked parents to complete a structured questionnaire about their experiences with the procedure at the follow-up visits (including potential problems, and satisfaction measured by a visual analogue scale from 0 - 100%). We defined highly or completely satisfied as a score of 90% or greater. We asked whether parents would be likely to choose NMC for a future son and how likely parents would be to recommend the procedure to a relative or a friend who had a baby boy.

SECONDARY OUTCOMES:
Staff impressions of the comparative safety, tolerability, and ease of use of the techniques (Mogen Clamp and Plastibell only). | After 4 months
  After all participant follow-up visits were completed, study staff were asked to fill-out a short semi-structured questionnaire of their subjective impressions of the two devices (Mogen Clamp and Plastibell only).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M. Plank, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Botswana-Harvard Partnership, Gaborone, Mochudi, Molepolole and Lobatse, Botswana

REFERENCES:
- See also: The Clearinghouse exists to expand global access to information and resources on male circumcision for HIV prevention. — http://www.malecircumcision.org/